CLINICAL TRIAL: NCT00791466
Title: Iodine Supplementation in Pregnant Women Living in Mild-to-moderately Iodine Deficient Areas in India and Thailand: Effects on Pregnancy Outcome and Infant Development
Brief Title: Maternal Iodine Supplementation and Effects on Thyroid Function and Child Development
Acronym: MITCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: St. John's Research Institute (Other); Mahidol University (Other); Unilever R&D (Industry); Swiss National Science Foundation (Other); Nestlé Foundation (Other)
Responsible Party: Principal Investigator, Alida Melse, Dr., Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MITCH-01
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Iodine Deficiency; Infant Development
Keywords: Iodine deficiency; Pregnancy; Thyroid function; Infant development; Growth
MeSH Terms: interventions — Iodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: Iodine
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Daily placebo supplementation from enrolment <14 wk of gestation until delivery
  Arms: 2
Dietary Supplement: Iodine — Daily supplementation with 200 µg iodine from enrolment <14 wk of gestation until delivery
  Arms: 1

SUMMARY:
Rationale: In regions of severe endemic goiter, the adverse effects of in utero iodine deficiency on neuromotor development are well established: randomized controlled trials of iodine supplements given to iodine deficient mothers before pregnancy or during early pregnancy improve motor and cognitive performance of their offspring. However, the potential adverse effects of mild-to-moderate iodine deficiency during pregnancy are unclear. Inadequate thyroid function in the fetus and newborn are the likely cause of brain damage in iodine deficiency.

Objective: To determine whether the daily oral administration of 200 µg iodine to pregnant women in areas of mild-to-moderate iodine deficiency improves maternal and newborn thyroid function, pregnancy outcome, birth weight, infant growth and cognitive performance.

Study design: Double-blind randomized controlled multicentre trial. Study population: Pregnant women (18-40 years) presenting at the clinic for their first prenatal visit will be recruited at two research sites, namely St. Martha's hospital in Bangalore, India and Ramathibodi Hospital, Mahidol University, Bangkok, Thailand. At each site, 400 women will be recruited.

Intervention: Half of the women will be randomized to iodine treatment (200 µg per day) and the other half to placebo throughout pregnancy.

Main study parameters/endpoints: Differences between group means in indicators of thyroid function, birth outcome, urinary iodine, breast milk iodine, infant growth, and psychomotor development.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years;
* Gestational age: ≤ 14 weeks (as judged by the date of the last menstrual period);
* Single pregnancy;
* Non-lactating;
* Planned residence in the area for the duration of the study (3 years).

Exclusion Criteria:

* TSH levels outside the normal range
* History of serious medical conditions such as HIV, hypertension, diabetes, renal, hepatic or cardiovascular disease, thyroid disorders, mental disorders;
* Use of iodine supplement.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 829 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Current primary outcome: Infant cognitive and motor development | Regular intervals up till 6 years of age
Original primary outcome: Maternal thyroid function | 3-month intervals during pregnancy, at delivery

SECONDARY OUTCOMES:
Birth outcome | At delivery
Maternal and infant urinary iodine | Regular intervals during pregnancy up till 2 years after delivery
Breast milk iodine | 3 and 6 months after delivery
Long-term follow up | Child age 2-6 years
  Anthropometrics, urinary iodine, thyroid hormones, WPPS, BRIEF-P, hearing thresholds

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, Prof. dr., Principal Investigator — Wageningen University; Alida Melse-Boonstra, PhD, Principal Investigator — Wageningen University
Locations (2):
- St. Johns Medical College and Research Institute, Bangalore, India
- Insitute of Nutrition, Mahidol University (INMU), Bangkok, Thailand

REFERENCES:
- [Background] Melse-Boonstra A, Gowachirapant S, Jaiswal N, Winichagoon P, Srinivasan K, Zimmermann MB. Iodine supplementation in pregnancy and its effect on child cognition. J Trace Elem Med Biol. 2012 Jun;26(2-3):134-6. doi: 10.1016/j.jtemb.2012.03.005. Epub 2012 May 8. PMID 22575544
- [Background] Gowachirapant S, Melse-Boonstra A, Winichagoon P, Zimmermann MB. Overweight increases risk of first trimester hypothyroxinaemia in iodine-deficient pregnant women. Matern Child Nutr. 2014 Jan;10(1):61-71. doi: 10.1111/mcn.12040. Epub 2013 Aug 13. PMID 23937433
- [Background] Jaiswal N, Melse-Boonstra A, Thomas T, Basavaraj C, Sharma SK, Srinivasan K, Zimmermann MB. High prevalence of maternal hypothyroidism despite adequate iodine status in Indian pregnant women in the first trimester. Thyroid. 2014 Sep;24(9):1419-29. doi: 10.1089/thy.2014.0071. Epub 2014 Jul 21. PMID 24923842
- [Background] Gowachirapant S, Jaiswal N, Melse-Boonstra A, Galetti V, Stinca S, Mackenzie I, Thomas S, Thomas T, Winichagoon P, Srinivasan K, Zimmermann MB. Effect of iodine supplementation in pregnant women on child neurodevelopment: a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2017 Nov;5(11):853-863. doi: 10.1016/S2213-8587(17)30332-7. Epub 2017 Oct 10. PMID 29030199
- [Background] Verhagen NJE, Gowachirapant S, Winichagoon P, Andersson M, Melse-Boonstra A, Zimmermann MB. Iodine Supplementation in Mildly Iodine-Deficient Pregnant Women Does Not Improve Maternal Thyroid Function or Child Development: A Secondary Analysis of a Randomized Controlled Trial. Front Endocrinol (Lausanne). 2020 Oct 6;11:572984. doi: 10.3389/fendo.2020.572984. eCollection 2020. PMID 33123091